CLINICAL TRIAL: NCT06666153
Title: A Clinical Study Evaluating the Safety, Tolerability, and Initial Efficacy of Therapeutic Immunological Agent for EBV Lymphoproliferative Diseases
Brief Title: Clinical Study of Therapeutic Immunological Agent for EBV Lymphoproliferative Diseases
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-68
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: CAEBV (Chronic Active Epstein-Barr Virus Infection) Syndrome; PTLDs
Keywords: EBV; immunotherapy; Lymphoproliferative disease, LPD; chronic active Epstein-Barr virus disease，CAEBV; Post-transplant lymphoproliferative disorders，PTLD
MeSH Terms: conditions — Syndrome; Lymphoproliferative Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Cohort (Experimental): EBV immunological agent administration on day 0,7,14,21 and 42 for Intradermal or Subcutaneous Injection
  Interventions: Biological: EBV immunological agent

INTERVENTIONS:
Biological: EBV immunological agent — 27 participants with will be enrolled in the study and divided into three groups, including EBV-LPD (Adults group), EBV-LPD (Children group) and PTLD (Adults group） each with 9 people.The participants will be divided into three different dose groups, and a "3+3" dose escalation design is used. The low dose is 5.0×10^5, the medium dose is 2.0×10^6 and the high dose is 5.0×10^6 for children and low dose is 5.0×10^6, the medium dose is 2.0×10^7 and the high dose is 5.0×10^7 for adults. Only one dose will be administered to each participant with EBV immunological agent combined with Toripalimab 240mg.

SUMMARY:
This study intends to conduct a prospective single-center open single-arm multi-dose escalation study on therapeutic immunological agent treatment in patients with Lymphoproliferative disease associated with EBV to observe the safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. For CAEBV patients and others with EBV-LPD 1). Patients who have signed informed consent before the trial and have a full understanding of the trial content, process and possible adverse reactions, and can complete the study according to the requirements of the trial protocol; 2). Patients with evidence consistent with the following diagnoses:

   a. Patients with the 2016 version of WHO's CAEBV diagnostic criteria (except

   B-lymphocyte involvement only) :
   * Persistent or recurrent infectious IM-like symptoms lasting for more than 3 months;

     * Increased EBV-DNA load in peripheral blood or tissue lesions: the level of EBV-DNA in peripheral blood was higher than 10^2.5 copies/μg DNA; ③ EBV-infected T cells or NK cells were found in the affected tissues or peripheral blood;

       ④ Exclude other possible diagnoses, such as primary EBV infection (IM), autoimmune diseases, neoplastic diseases, other viral infections (HBV, HIV, HCV, etc.), and congenital or secondary immunodeficiency diseases; Or b. EBV-PLD patients with evidence consistent with pathological diagnosis of EBV antigen positive; 3). Male and female, 2-70 years old (including the critical value); 4). Patients with EBV-DNA≥1000 copies/mL or EBER+; 5). Before the study, total bilirubin ≤ 2 times of the upper limit of normal value, blood creatinine ≤ 1.5 times of normal value; Fibrinogen can be corrected to ≥0.6g/L after infusion.

       6). Before the study, hemoglobin ≥60g/L, platelets ≥50×10^9/L, neutrophil count ≥1×10^9/L; 7). Echocardiography showed LVEF ≥ 50%; 8). Women of childbearing age must confirm through a pregnancy test that they are not pregnant and be willing to use effective contraception during the test period and for ≥12 months after the last dose; 9). The compliance was good, and the patients and their families were willing to cooperate with the later follow-up.
2. For PTLD patients 1). Patients who have signed informed consent before the trial and have a full understanding of the trial content, process and possible adverse reactions, and can complete the study according to the requirements of the trial protocol; 2). Patients diagnosed with PTLD WHO have received SOT or HSCT (refer to WHO 2016 diagnostic criteria); 3). Male and female, 18-70 years old (including the critical value); 4). Patients with EBV-DNA≥1000 copies/mL or EBER+; 5). Women of childbearing age must confirm through a pregnancy test that they are not pregnant and be willing to use effective contraception during the test period and for ≥12 months after the last dose; 6). Good compliance, patients and their families are willing to cooperate with later follow-up.

Exclusion Criteria:

Patients were excluded if they met any of the following criteria:

1. For CAEBV patients and others with EBV-LPD 1). Participated in other drug clinical trials within 4 weeks; 2). Pregnant or lactating patients; 3). Patients with severe heart, lung and kidney diseases; 4). Active gastrointestinal bleeding; 5). The patient has active pulmonary tuberculosis, bacterial or fungal infection (≥ Grade 2 of NCI-CTC, 3rd edition); Have a history of herpes simplex, herpes zoster or chickenpox within 3 months; 6). People with a history of psychotropic drug abuse and unable to quit or patients with mental disorders; 7). The subject has any active autoimmune disease or history of autoimmune disease; 8). In the judgment of the investigator, there is a serious concomitant disease that endangers the patient's safety or interferes with the patient's completion of the study.
2. For PTLD patients 1). Patients with active aGVHD III-IV and/or mild and severe cGVHD; 2). Had received other cellular immunotherapy clinical studies 30 days before enrollment; 3). Pregnant or lactating patients; 4). Intracranial hypertension or confusion; Respiratory failure; Patients with diffuse intravascular coagulation; 5). Organ failure patients: (1) Heart :NYHA level IV cardiac function; (2) Liver: Grade C, reaching the Child-Turcotte liver function grade; (3) Kidney: renal failure, uremia; (4) Lungs: symptoms of respiratory failure. 6). Patients with active gastrointestinal bleeding; 7). Patients with severe non-compensatory hypertension; 8). Patients with severe non-compensatory diabetes; 9). The patient has active pulmonary tuberculosis, bacterial or fungal infection (≥ Grade 2 of NCI-CTC, 3rd edition); Have a history of herpes simplex, herpes zoster or chickenpox within 3 months; 10). Those who have a history of psychotropic drug abuse and cannot quit or those with mental disorders; 11). The subject has any active autoimmune disease or history of autoimmune disease; 12). Other possible diagnoses, such as primary EBV infection (IM), neoplastic diseases, other viral infections (HBV, HIV, HCV, etc.), and congenital or secondary immunodeficiency diseases; 13). According to the judgment of the investigator, there is a serious harm to the safety of the patient or affect the completion of the study.

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | up to 12 months
  Number of participants who experience grade 1 or higher adverse events, as defined by Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0).

SECONDARY OUTCOMES:
Quality of life for patients | up to 12 months
  The EORTC QLQ-C30 consists of five functional scales, nine symptom scales and one global quality of life (QoL) scale, and has been validated in an international setting
Effectiveness | up to 12 months
  The number of subjects with CR and PR, calculate the duration from the time of initial administration to the date of disease progression or the date of subject's death

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Clerico M, Dogliotti I, Aroldi A, Consoli C, Giaccone L, Bruno B, Cavallo F. Post-Transplant Lymphoproliferative Disease (PTLD) after Allogeneic Hematopoietic Stem Cell Transplantation: Biology and Treatment Options. J Clin Med. 2022 Dec 19;11(24):7542. doi: 10.3390/jcm11247542. PMID 36556158
- [Result] Hartlage AS, Liu T, Patton JT, Garman SL, Zhang X, Kurt H, Lozanski G, Lustberg ME, Caligiuri MA, Baiocchi RA. The Epstein-Barr Virus Lytic Protein BZLF1 as a Candidate Target Antigen for Vaccine Development. Cancer Immunol Res. 2015 Jul;3(7):787-94. doi: 10.1158/2326-6066.CIR-14-0242. Epub 2015 Mar 3. PMID 25735952
- [Result] Savoldo B, Huls MH, Liu Z, Okamura T, Volk HD, Reinke P, Sabat R, Babel N, Jones JF, Webster-Cyriaque J, Gee AP, Brenner MK, Heslop HE, Rooney CM. Autologous Epstein-Barr virus (EBV)-specific cytotoxic T cells for the treatment of persistent active EBV infection. Blood. 2002 Dec 1;100(12):4059-66. doi: 10.1182/blood-2002-01-0039. Epub 2002 Aug 1. PMID 12393655
- [Result] Bollard CM, Gottschalk S, Helen Huls M, Leen AM, Gee AP, Rooney CM. Good manufacturing practice-grade cytotoxic T lymphocytes specific for latent membrane proteins (LMP)-1 and LMP2 for patients with Epstein-Barr virus-associated lymphoma. Cytotherapy. 2011 May;13(5):518-22. doi: 10.3109/14653249.2011.561983. Epub 2011 Mar 1. No abstract available. PMID 21361747
- [Result] Ma Y, Zhang P, Bao Y, Luo H, Wang J, Huang L, Zheng M. Outcomes of programmed death protein-1 inhibitors treatment of chronic active Epstein Barr virus infection: A single center retrospective analysis. Front Immunol. 2023 Mar 10;14:1093719. doi: 10.3389/fimmu.2023.1093719. eCollection 2023. PMID 36969150
- [Result] Song Y, Wang J, Wang Y, Wang Z. Ruxolitinib in Patients With Chronic Active Epstein-Barr Virus Infection: A Retrospective, Single-Center Study. Front Pharmacol. 2021 Sep 6;12:710400. doi: 10.3389/fphar.2021.710400. eCollection 2021. PMID 34552486
- [Result] Hui KF, Cheung AK, Choi CK, Yeung PL, Middeldorp JM, Lung ML, Tsao SW, Chiang AK. Inhibition of class I histone deacetylases by romidepsin potently induces Epstein-Barr virus lytic cycle and mediates enhanced cell death with ganciclovir. Int J Cancer. 2016 Jan 1;138(1):125-36. doi: 10.1002/ijc.29698. Epub 2015 Aug 11. PMID 26205347
- [Result] Al-Mansour Z, Nelson BP, Evens AM. Post-transplant lymphoproliferative disease (PTLD): risk factors, diagnosis, and current treatment strategies. Curr Hematol Malig Rep. 2013 Sep;8(3):173-83. doi: 10.1007/s11899-013-0162-5. PMID 23737188
- [Result] Kawa K, Sawada A, Sato M, Okamura T, Sakata N, Kondo O, Kimoto T, Yamada K, Tokimasa S, Yasui M, Inoue M. Excellent outcome of allogeneic hematopoietic SCT with reduced-intensity conditioning for the treatment of chronic active EBV infection. Bone Marrow Transplant. 2011 Jan;46(1):77-83. doi: 10.1038/bmt.2010.122. Epub 2010 May 24. PMID 20498651
- [Result] Sawada A, Inoue M, Kawa K. How we treat chronic active Epstein-Barr virus infection. Int J Hematol. 2017 Apr;105(4):406-418. doi: 10.1007/s12185-017-2192-6. Epub 2017 Feb 16. PMID 28210942
- [Result] Lu G, Xie ZD, Zhao SY, Ye LJ, Wu RH, Liu CY, Yang S, Jin YK, Shen KL. Clinical analysis and follow-up study of chronic active Epstein-Barr virus infection in 53 pediatric cases. Chin Med J (Engl). 2009 Feb 5;122(3):262-6. PMID 19236801
- [Result] Kimura H, Morishima T, Kanegane H, Ohga S, Hoshino Y, Maeda A, Imai S, Okano M, Morio T, Yokota S, Tsuchiya S, Yachie A, Imashuku S, Kawa K, Wakiguchi H; Japanese Association for Research on Epstein-Barr Virus and Related Diseases. Prognostic factors for chronic active Epstein-Barr virus infection. J Infect Dis. 2003 Feb 15;187(4):527-33. doi: 10.1086/367988. Epub 2003 Jan 28. PMID 12599068
- [Result] Yonese I, Sakashita C, Imadome KI, Kobayashi T, Yamamoto M, Sawada A, Ito Y, Fukuhara N, Hirose A, Takeda Y, Makita M, Endo T, Kimura SI, Ishimura M, Miura O, Ohga S, Kimura H, Fujiwara S, Arai A. Nationwide survey of systemic chronic active EBV infection in Japan in accordance with the new WHO classification. Blood Adv. 2020 Jul 14;4(13):2918-2926. doi: 10.1182/bloodadvances.2020001451. PMID 32598475
- [Result] Kimura H, Hoshino Y, Kanegane H, Tsuge I, Okamura T, Kawa K, Morishima T. Clinical and virologic characteristics of chronic active Epstein-Barr virus infection. Blood. 2001 Jul 15;98(2):280-6. doi: 10.1182/blood.v98.2.280. PMID 11435294